CLINICAL TRIAL: NCT06703541
Title: Duke/UNC Alzheimer's Disease Center Clinical Cohort
Brief Title: ADRC Clinical Cohort (Alzheimer's Disease)
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00103958; 1P30AG072958 (NIH)
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment; Dementia
Keywords: Genetic risk; Alzheimer Disease; Dementia; Aging; Alzheimer's Disease Research Center (ADRC)
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine, and cerebrospinal fluid samples will be obtained and stored.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Participants aged 25-44: Subjects ages 25 to 44 at enrollment with normal cognition will undergo baseline visits including:
  * Demographics
  * Family history, medical history, current medications
  * General physical and neurological exam, sensory and motor testing
  * Vital signs
  * Blood sample collected for PT/INR, blood count, genetic testing, and storage for future unspecified research on cognition and disorders associated with altered cognition
  * Urine sample
  * Neuropsychological testing
  * Retinal imaging
  * Testing of memory, thought processes, and recognition
  * MRI
  * Lumbar puncture
- Participants aged 45-80: Subjects ages 45 to 80 at enrollment with normal cognition, mild cognitive impairment, or dementia will undergo baseline visits including:
  * Demographics and project partner demographics
  * Family history, medical history, current medications
  * General physical and neurological exam, sensory and motor testing
  * Vital signs
  * Blood sample collected for PT/INR, blood count, genetic testing, and storage for future unspecified research on cognition and disorders associated with altered cognition
  * Urine sample
  * Neuropsychological testing
  * Retinal imaging
  * Testing of memory, thought processes, and recognition
  * MRI
  * Lumbar puncture
  Participants will be asked to participate in yearly evaluations until the time of death. Participants can withdraw at any time.

SUMMARY:
The purpose of the study is to establish a clinical cohort for the Duke/UNC Alzheimer's Disease Research Center (ADRC). The cohort will be composed of subjects ages 25 to 44 at enrollment with normal cognition and subjects ages 45 to 80 at enrollment with normal cognition, mild cognitive impairment, or a dementia diagnosis. Initial data including demographics, medical and family history, physical exam, and neuropsychological testing will be obtained. Participants will be asked to contribute a blood sample, a urine sample, a cerebrospinal fluid sample, and undergo a MRI scan. The cohort ages 45 to 80 will be seen yearly until death to evaluate medical status, undergo neuropsychological testing and possibly collect additional samples or undergo additional imaging. All data will be de-identified and stored by the ADRC.

The purpose of this study is to examine normal cognition, mild cognitive impairment and Alzheimer's disease and related dementias (ADRD) as people get older. The investigators also hope to be able to assess risk factor information of the role of genes and environmental exposures (for example health conditions, diet, and medications) in Alzheimer's disease and related disorders (ADRD) and other conditions of aging.

The biological samples collected in the study will create a repository. A repository is a collection of blood and tissue samples from people with certain diseases and conditions. For the purpose of this research, the investigators hope to help researchers learn more about Alzheimer's disease and related disorders and other conditions of aging.

DETAILED DESCRIPTION:
The purpose of the study is to build a clinical cohort of adult research subjects with normal cognition, mild cognitive impairment (MCI), and dementia due to Alzheimer's disease and other related dementias (ADRD), enrolling 100 subjects per year. The primary objective of this cohort will be to advance research on neurodegenerative brain disorders and the role of age, sex and genetics (especially APOE genotype) on their manifestation.

The primary objective is to create a clinical cohort for the Duke/UNC Alzheimer's Disease Research Center (ADRC). The ages of the cohort will be 25 to 44 and 45 to 80 at the time of enrollment. Subjects aged 45 to 80 must have a project partner as part of the study. The cohort will undergo baseline data collection according to the Uniform Data Set, version 3 set forth by the National Alzheimer's Coordinating Center including medical and family history, physical exam, neuropsychological testing, blood and urine sample, cerebrospinal fluid sample, and brain MRI. A subject's project partner can be substituted for another one, and if so, the new potential project partner will be consented into the study. Subjects in the ages 45 to 80 group will be re-evaluated every year with a medical history update, physical exam, and neuropsychological testing.

Additional blood, fluid or imaging may be requested at later dates. As part of their enrollment in the cohort the subjects will be presented yearly to a consensus committee to confirm diagnosis. A subset of the cohort ages 45 to 80, unable or unwilling to have the Lumbar Puncture, may alternately be offered to supplement a PET Scan to confirm diagnosis if/when AD symptoms are present.

The Duke/UNC ADRC obtained funding from the National Institute of Aging (NIA) in September 2021 and is an NIA designated ADRC program.

Subjects with normal cognition, mild cognitive impairment and dementia diagnosis will be recruited from clinical visits at the Duke Neurology Memory Disorders Clinic at Morreene Road. Subjects will also be enrolled by self-referral and active recruitment through participation in existing studies, registries, educational talks at community organizations and community health fairs. Subjects in the ages 45-80 cohort must have a dedicated project partner of their choice at time of enrollment. The project partner is an individual who knows the participant well, preferably a family member (e.g. spouse, adult child).

Written informed consent will be obtained from all participants and their project partners (via paper or via eConsent).

Subjects will have an initial visit with information/history gathering, physical exam, neuropsychological testing, and blood draw. The project partner will be asked questions about the participant's activities of daily living (ADLs), mood, and day to day behaviors. Subjects will have follow-up visits coordinating imaging, lumbar puncture, and donation of other biological samples.

A subset of the total age 45 to 80 cohort (up to 100 total subjects), unable or unwilling to have the Lumbar Puncture, may alternately be offered to supplement a PET Scan to confirm diagnosis if/when Alzheimer's Disease symptoms are present.

Subjects and project partners in the age 45 to 80 cohort will have an annual follow-up visit as long as they can participate, preferably in person, but may also occur over the telephone if necessary.

All information gathered at the initial visit and annual follow-up will be entered into the Uniform Data Set (UDS), version 3, a longitudinal data set that is submitted to the National Alzheimer's Coordinating Center (NACC). At baseline and at yearly follow-up, a consensus committee will meet to make a diagnosis based on history and presentation, neuropsychological testing, imaging, and biomarker information.

All activities are research-related. Subjects ages 25 to 44 and ages 45 to 80 will have the following visit schedule:

Baseline Visits (typically over 3 visits, completed within 60 days of initial visit):

* Informed consent will be obtained from subject and project partner
* Subjects will be assigned a coded research identification number
* Demographics and project partner demographics
* Family history, medical history and current medications
* General physical and neurological exam, including sensory and motor testing
* Vital signs
* Blood sample will be collected for PT/INR, blood count, genetic testing, and storage at Duke for future unspecified research on cognition and disorders associated with altered cognition
* Laboratory test results will be reviewed for normal PT/INR and blood count before scheduling the lumbar puncture
* Urine sample
* Neuropsychological testing
* Retinal imaging (non-invasive screening of subject's eyes to look for potential signs of Alzheimer's or related disorders)
* Additional testing of subject's memory, thought processes, and recognition
* MRI
* Lumbar puncture

Yearly evaluations:

- Subjects and project partners in the ages 45 to 80 cohort will be contacted approximately every 12 months for a follow-up evaluation. At the yearly follow up evaluation the investigators will update medical information and perform neuropsychological testing. The investigators may also collect additional blood or CSF and additional imaging. These follow-up evaluations are done ideally in person but also can be conducted over the telephone. Participants will be asked to participate in yearly evaluations until the time of death. Participants can withdraw from the study at any time without concern for the future of their care.

Consensus Committee Diagnosis:

After data collection is completed, a consensus committee composed of representatives from neurology, neuropsychology, and imaging will meet on a bi-weekly to monthly basis to review information on each subject and come to a consensus diagnosis. Each subject will be reviewed at baseline and yearly.

Storage of samples:

Blood and CSF samples will be stored. Samples will not contain any PHI and will be assigned a Repository ID number. Study staff will maintain the link between the PHI and samples.Samples will be stored indefinitely or until samples are exhausted. Subjects can request to have their samples withdrawn by sending a written request to the PI.

Research and Specimen Sharing:

The investigators will share subject's coded biological samples and data with the National Cell Repository for Alzheimer's Disease and Related Dementias (NCRAD), a research facility at Indiana University that is supported by the National Institute on Aging to facilitate genetic research in Alzheimer disease, aging, and related disorders.

All biological samples sent to NCRAD will also be stored indefinitely and processed at NCRAD for use by qualified scientists at other Alzheimer's Disease Centers and other research centers (including other academic and commercial laboratories studying Alzheimer's disease, aging, and other related disorders). In addition to the blood sample, some coded demographic information about the subject (age/year of birth, family history of dementia, and diagnosis) will be sent to NCRAD. Subject identity will not be shared with NCRAD or with any other outside investigators.

External investigators wishing to gain access to these data and/or samples will be required to submit a separate IRB application and consent for this purpose. All proposals must be internally reviewed to assure appropriate use of the data/specimens and to determine feasibility and availability of resources. All requests and approvals for usage are tracked internally. The investigators also request copies of any publications from all investigators that resulted from, or included, data/specimens from our database/repository.

It must be emphasized that all data/specimens released from the Duke ADRC database/repository are deidentified. All data/specimens are coded by a unique Duke ADRC ID number rather than by name. Data and specimen information are maintained in the database according to identifier number and not by name.

The database/repository will be maintained indefinitely as long as funding is available or until the data/specimens are exhausted.

ELIGIBILITY:
Inclusion Criteria:

* Each subject must be ≥ 25 to ≤ 80 years of age.
* Each subject must be able to read at a 6th grade level, as determined by the investigator, and must have a history of academic achievement and/or employment sufficient to exclude intellectual disability.
* Each subject (or legal representative) must sign the informed consent form after the scope and nature of the investigation have been explained to them, and before screening assessments. Some consent may be obtained via phone script and REDCap eConsent.
* Each participant must be willing to have an MRI and a lumbar puncture, or alternately (to the lumbar puncture) a series of PET scans.
* Each participant ages 45 to 80 must have a study partner who agrees to participate in the study and who is able to read at a 6th grade level, as determined by the investigator, and must have a history of academic achievement and/or employment sufficient to exclude intellectual disability.

Exclusion Criteria:

* Evidence of a clinically relevant or unstable neurological disorder including history of multiple head injuries, stroke or other CNS conditions (MS, Parkinson's disease, etc.)
* Evidence of a clinically relevant or unstable psychiatric disorder.
* History of alcoholism or drug dependency/abuse within the last 2 years before enrollment.
* GAD-7 score >9 and/or PHQ-8 score >9
* An ongoing uncontrolled, clinically significant medical condition such that, in the judgment of the investigator, a subject's participation in the trial would pose a significant medical risk to the subject.
* Contraindication or intolerance to 3T MRI investigations, including implanted devices
* History of malignancy of any organ system, treated or untreated, within the past 60 months, regardless of whether there is evidence of local recurrence or metastases. However localized nonmalignant tumors not requiring systemic chemo- or radiotherapy, localized basal or squamous cell carcinoma of the skin, or in-situ cervical cancer are permitted.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals aged 25 to 44 at enrollment with normal cognition, and individuals aged 45 to 80 at enrollment with normal cognition, mild cognitive impairment, or a dementia diagnosis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-07-21 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants enrolled who are aged 25 to 44 with normal cognition | Until the end of the study, approximately 5 years
  The primary objective of this cohort will be to advance research on neurodegenerative brain disorders and the role of age, sex and genetics (especially APOE genotype) on their manifestation.
Number of participants enrolled who are aged 45 to 80 with normal cognition | Until the end of the study, approximately 5 years
  The primary objective of this cohort will be to advance research on neurodegenerative brain disorders and the role of age, sex and genetics (especially APOE genotype) on their manifestation.
Number of participants enrolled who are aged 45 to 80 with mild cognitive impairment (MCI) | Until the end of the study, approximately 5 years
  The primary objective of this cohort will be to advance research on neurodegenerative brain disorders and the role of age, sex and genetics (especially APOE genotype) on their manifestation.
Number of participants enrolled who are aged 45 to 80 with dementia | Until the end of the study, approximately 5 years
  The primary objective of this cohort will be to advance research on neurodegenerative brain disorders and the role of age, sex and genetics (especially APOE genotype) on their manifestation.

CONTACTS AND LOCATIONS:
Overall Officials: Heather E Whitson, MD, MHS, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Duke/UNC Alzheimer's Disease Research Center website — https://dukeuncadrc.org/

DOCUMENTS (2):
  • Study Protocol (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT06703541/Prot_002.pdf
  • Informed Consent Form (2025-08-14): https://cdn.clinicaltrials.gov/large-docs/41/NCT06703541/ICF_003.pdf